CLINICAL TRIAL: NCT01023737
Title: Inhibition of Autophagy in Solid Tumors: A Phase I Pharmacokinetic and Pharmacodynamic Study of Hydroxychloroquine in Combination With the HDAC Inhibitor Vorinostat for the Treatment of Patients With Advanced Solid Tumors With an Expansion Study in Advanced Renal and Colorectal Cancer
Brief Title: Hydroxychloroquine + Vorinostat in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDD 08-52; 08-462H (Other: UT Health San Antonio)
Record Dates: First submitted 2009-07-22; First posted 2009-12-02 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Malignant Solid Tumour
Keywords: Malignant Solid Tumor; Solid Tumor; Hydroxychloroquine; Vorinostat
MeSH Terms: interventions — Hydroxychloroquine; Vorinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxychloroquine and Vorinostat (Experimental): Oral administration of Vorinostat will be begin on Cycle 1 Day 1 at 300mg and will be continued daily and HCQ will be administered starting on Day 2 of Cycle 1 and both will be continued daily thereafter until progression of disease or unacceptable toxicity develops.
  Interventions: Drug: Hydroxychloroquine; Drug: Vorinostat

INTERVENTIONS:
Drug: Hydroxychloroquine — The HCQ study dose levels are defined as 400mg/day, 600mg/day, 800mg/day and 1000mg/day (oral dosing)during the phase I MTD determination. HCQ will be administered starting on Day 2 of Cycle 1 and will be continued daily thereafter until progression of disease or unacceptable toxicity develops.
  Other Names: HCQ
Drug: Vorinostat — Oral administration of Vorinostat will be begin on Cycle 1 Day 1 at 300mg and will be continued daily thereafter until progression of disease or unacceptable toxicity develops.
  Other Names: Suberoylanilide Hydroxamic Acid

SUMMARY:
This study is an open label non randomized study of hydroxychloroquine (HCQ) with histone deacetylase (HDAC) inhibitor Vorinostat in patients with advanced solid tumors to determine the maximum tolerated dose (MTD) and to evaluate the safety and antitumor activity of this drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 16 years of age
* Patients must have a histologically confirmed non-hematological malignancy. Patients must have received and failed standard treatment for their malignancy; patients for whom no standard treatment is available will also be eligible.
* Patients must have an ECOG PS at 0, 1, or 2
* Patients must have adequate hematologic, renal and liver function (i.e. absolute Neutrophil count > 1000/mm3, platelets > 75,000/mm3); creatinine

  * 2 times the upper limits of normal (ULN) total bilirubin ≤ 1.5 mg/dl, ALT and AST £ 3 times above the upper limits of the institutional norm ALT, AST can be < 5 times upper limits of normal if patients have hepatic involvement.
* Patients must be able to provide written informed consent.
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception. Women of childbearing potential must have a negative pregnancy test. The anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant.
* Complete supportive and palliative care will continue to be provided to ameliorate signs and symptoms that were pre-existing or may arise while on study and which do not interfere with the objectives of the study.
* Tumor blocks available from previous surgery/biopsy.

At the tumor specific expansion, only patients with metastatic colorectal and renal cell cancers will be enrolled. Patients with metastatic colorectal and renal cancer must have been treated and progressed or intolerant to standard care therapy.

Patients with colorectal cancer must been treated in the past with Irinotecan and/or Oxaliplatin and/or AvastinIEGFR therapy or intolerant to these agents. No more than 4 lines of therapy permitted in the metastatic setting. Patients with colorectal cancer may enroll irrespective of K-Ras mutational status, although this will be documented.

Patients with renal cell cancer must have been treated with a VEGF targeted therapy and/or mTOR inhibitor. No more than 4 lines of therapy permitted in the metastatic setting.

Prior treatment with Vorinostat and HCQ are not permitted in each tumor type.

Exclusion Criteria:

* Patients with uncontrolled brain metastases.
* Due to risk of disease exacerbation patients with porphyria are not eligible.
* Due to risk of disease exacerbation patients with psoriasis are ineligible unless the disease is well controlled and they are under the care of a specialist for the disorder who agrees to monitor the patient for exacerbations.
* Patients with previously documented macular degeneration or diabetic retinopathy.
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for Nitrosoureas or Mitomycin C) prior to entering the study or those who have not recovered from adverse events to ≤ grade 1 due to agents administered more than 4 weeks earlier. For targeted therapies patients will need to clear for 5 half lives.
* Patients may not be receiving any other investigational agents.
* Patients should not have taken valproic acid or another histone deacetylase inhibitor for at least 2 weeks prior to enrollment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat or HCQ.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Major surgery or significant traumatic injury occurring within 21 days prior to treatment.
* Clinically significant hypercalcemia (including vomiting, dehydration and neurological symptoms).
* QTc > 500 ms at baseline (average of 3 determinations at 10 minutes interval).
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease. Patients with NJ, J or G tube will not be allowed to participate.
* Pregnant women are excluded from this study because SAHA has the potential for teratogenic or abortifacient effects
* Patients with known hepatitis B or C or HIV infection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-11; Primary Completion 2017-12-05 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of Hydroxychloroquine (HCQ) in combination with Vorinostat in patients with advanced solid tumors | 6+ months, MTD is assessed during the 1st cycle

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of HCQ in combination with Vorinostat in this patient population as determined by toxicity profile, incidence and rating according to NCI/CTC v3.0 criteria. | 1 year
To evaluate the antitumor activity of HCQ in combination with Vorinostat as determined by response rate and progression free survival (exploratory) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sukeshi Patel Arora, MD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Cancer Therapy & Research Center University of Texas Health Science Center San Antonio, San Antonio, Texas, United States